CLINICAL TRIAL: NCT05107947
Title: Light in Frail Elderly - the Effect of a Dynamic Light for Sleep and Circadian Rhythm
Acronym: LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-02765
Record Dates: First submitted 2021-10-26; First posted 2021-11-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Aged; Circadian Rhythm; Cognition; Fatigue; Humans; Light; Melatonin; Sleep; Biocentric; Frailty; Karolinska Sleepiness Score; Inflammation
MeSH Terms: conditions — Fatigue; Frailty; Inflammation

STUDY DESIGN:
Intervention Model Description: One intervention group and one control group
Masking Description: Interventions constitutes of a different lighting environment therefore not possible to mask.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention biocentric light environment (Experimental): In all study rooms, a biocentric lighting environment will be able to be created by activating a special lighting system. In these rooms, light will change dynamically both in spectral distribution and intensity during the day. During the day, color temperature and intensity are high (1000 lux and up to 6500 K) to decrease both intensity and color temperature during the evening.
  Interventions: Other: Biocentric light
- Control standard light environment (No Intervention): Standard static light environment.

INTERVENTIONS:
Other: Biocentric light — Light that changes in intensity and spectral distribution during the day to mimick daylight. High in intensity and high circadian stimulus during daytime and low intensity and low circadian stimulus during late afternoon and night.
  Arms: Intervention biocentric light environment

SUMMARY:
The aim of this project is to evaluate the effect of a dynamic light in order to improve the circadian rhythm, provide a better sleep and well-being, and in the long run an improved recovery. The primary question is whether dynamic artificial light with circadian stimulus can affect the circadian rhythm. The secondary question is whether this also provides better sleep and well-being.

The group that is particularly interesting to study is a geriatric population that is more sensitive to circadian rhythm disorders, sleep disorders and confusion in connection with hospitalization and that can be of particular benefit from this intervention.

DETAILED DESCRIPTION:
This is a randomized, prospective study where the diurnal variation of melatonin as well as sleep-related parameters (sleep duration and sleep quality) will be investigated with regards to light exposure during the hospital stay. Furthermore, it is investigated how psychological and cognitive functions are affected by light intervention and whether this is related to improved sleep or not. The study includes a total of 300 patients over the age of 65 who are cared for in an internal medicine or orthopedic surgery department at Skåne University Hospital in Malmö. The measurement period in the project is intended to be carried out during the period of October 2021-February 2022. Hospital rooms in the orthopedic department and in the medical department constitute the study environment. In all rooms, a biocentric lighting environment will be able to be created by activating a special lighting system. In these rooms, light will change dynamically both in spectral distribution and intensity during the day. During the day, color temperature and intensity are high (1000 lux and up to 6500 K) to decrease both intensity and color temperature during the evening. By weighing together spectral distribution and brightness, the circadian stimulus of the light environment can be calculated. The biocentric light provides a light with a high circadian stimulus during the morning and early afternoon. The biocentric light can be turned on (intervention) or off (control). When control setting, the standard normal light constitutes the light environment.

In all rooms included in the study, an accurate measurement of light conditions is carried out both with regard to spectral distribution and light intensity. Furthermore, patients will carry light meters to measure the actual amount of light to which patients are exposed. The study includes two arms, an intervention group and a control group. Patients who are assigned to one of the study rooms, and meet the inclusion criteria, will be asked to participate in the study. Patients are randomized to activate the biocentric light environment or standard light environment. The patients who are cared for in a biocentric light environment are included in the intervention group and those who are cared for in rooms with a standard light environment are included in the control group.

300 patients are to be included in the study. Surveys concerning alertness, sleep will be carried out. The frailty and a rapid test for delirium will be assessed. The patients will wear an actiwatch that records their sleep. For a small group of patients, also saliva melatonin will be collected every 4th hour from 7 pm to 11 am for two different nights 3 days apart. The results will be compared between the patients in the intervention group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 65 years
* Admitted to one of the included study rooms

Exclusion Criteria:

* Overdose addictive substance
* Acute neurological disease
* Melatonin treatment
* Probable survival <5 days
* Severe visual impairment that makes reading impossible
* Age <65 years
* Inability to understand Swedish in speech and writing
* Inability to consent to participate in the study
* The patient is on any of the following medicines:

  * Medications for Parkinson's disease
  * Neuroleptics (including lithium)
  * Dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Melatonin curve | Change after three days of biocentric light exposure
  A change in the phase of the melatonin curve

SECONDARY OUTCOMES:
Sleep | Increased total sleep time after three days of biocentric light exposure
  Change in sleep time

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Selvander, MD, PhD, Principal Investigator — Lunds Universitet
Locations (1):
- Skåne University Hospital Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No